CLINICAL TRIAL: NCT01997580
Title: Phase 4 Study of Escitalopram Treatment and Biomarkers in Major Depressive Disorder
Brief Title: Electrophysiologic Parameters and Biomarkers Predicting Treatment Response in Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Jae Seung Chang, Associate Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: A121987
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: depression; treatment; electrophysiology; biomarker
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental): depressed patients receiving escitalopram treatment
  Interventions: Drug: escitalopram
- Control (No Intervention): healthy controls matched for age, gender, and BMI

INTERVENTIONS:
Drug: escitalopram — SSRI antidepressant
  Other Names: lexapro
  Arms: Escitalopram

SUMMARY:
To explore electrophysiologic parameters and biomarkers predicting treatment response of patients with major depressive disorder To explore electrophysiologic parameters and biomarkers predicting suicide risk of patients with major depressive disorder

DETAILED DESCRIPTION:
Case-control study Repeated measures design

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR major depressive disorder
* aged between 20 and 80
* durg-naive or drug-free

Exclusion Criteria:

* DSM-IV-TR substance-related disorders (except nicotine)
* significant medical or neurological conditions
* mental retardation or organic brain damage

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline frequency of maximum of cross-spectrum during 6 weeks (Hz) | 0, 3, 7, 14, and 42 days
  the link between the normalized high frequency component of heart rate variability (HRV-HFnu) representing cardiac vagal modulation and frontal alpha power related to resting state

SECONDARY OUTCOMES:
Change in cardiorespiratory coupling during 6 weeks | 0, 3, 7, 14, and 42 days
  change in value of cross-sample entropy measured by combining sample entropies of heart rate and respiration
Change in HF during 6 weeks | 0, 3, 7, 14, and 42 days
  change in high frequency component of heart rate variability
Change in persistent homology during 6 weeks | 0, 3, 7, 14, and 42 days
  change in disconnection pattern of EEG channel activities measured by Euclidean distance during 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jae Seung Chang, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Chang JS, Yoo CS, Yi SH, Her JY, Choi HM, Ha TH, Park T, Ha K. An integrative assessment of the psychophysiologic alterations in young women with recurrent major depressive disorder. Psychosom Med. 2012 Jun;74(5):495-500. doi: 10.1097/PSY.0b013e31824d0da0. Epub 2012 Mar 9. PMID 22408133
- See also: health information about depression — http://www.nlm.nih.gov/medlineplus/ency/article/000945.htm